CLINICAL TRIAL: NCT05059236
Title: Open-label Study of Androgen Receptor Inhibition With dArolutamide Plus Androgen Deprivation Therapy (ADT) Versus ADT in Men With Metastatic Hormone-Sensitive Prostate Cancer Using an External Control Arm
Brief Title: A Study to Learn How Well Darolutamide Administered Together With Androgen Deprivation Therapy (ADT) Works in Men With Metastatic Hormone-sensitive Prostate Cancer. Results Will be Compared With ADT Alone From a Previously Conducted Study.
Acronym: ARASEC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21516
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
Keywords: Metastatic hormone-sensitive prostate cancer (mHSPC); Prostate Cancer; Darolutamide; Nubeqa
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Darolutamide+ADT (Experimental): Participants will receive darolutamide plus ADT in the ARASEC treatment arm. The control arm for the study will be derived from the participants treated with ADT alone in the CHAARTED trial using a matching approach
  Interventions: Drug: Darolutamide (BAY1841788, Nubeqa); Other: ADT

INTERVENTIONS:
Drug: Darolutamide (BAY1841788, Nubeqa) — 300 mg per tablet, oral administration with food
Other: ADT — LHRH agonist/antagonist or orchiectomy

SUMMARY:
The purpose of the study is to assess if the addition of darolutamide to ADT compared with ADT alone would result in superior clinical efficacy in participants with metastatic hormone-sensitive prostate cancer (mHSPC) by progression-free survival.

The researchers want to learn how long it takes for the cancer to get worse (also known as "progression-free survival") by either increasing symptoms, new metastases, PSA rise or death. All participants will be on treatment and take darolutamide with ADT until their cancer spreads, they have a medical problem, or they leave the study. The results will then be compared with patients' results from another study who received ADT alone (CHAARTED).

This study will also assess safety by gathering adverse event information throughout the duration of the study. An adverse event is any medical problem, related or not to study treatment that a participant has during a study.

The study drug, darolutamide, is already available for doctors to prescribe to patients with prostate cancer that has not yet spread to other parts of the body. It works by blocking a protein called a receptor from attaching to a hormone called androgen that is found in men. This protein can also be found in prostate cancer cells. ADT is a treatment that doctors are currently able to prescribe to patients with mHSPC. ADT is used to lower the amount of the androgen hormone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate. Participants may have begun androgen-deprivation therapy (up to 120 days prior to enrollment). Note: Relugolix is not permitted as ADT in this study.
* Metastatic disease and will be stratified by presence of high volume or low volume disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1 or 2
* Adequate bone marrow, liver and renal function within 4 weeks of enrollment
* At least 4 weeks since prior major surgery and recovered from all toxicity from such surgery prior to enrollment
* Prior adjuvant or neoadjuvant hormonal therapy allowed provided the following criteria are met:

  * Therapy was discontinued ≥ 12 months ago AND there was a clinical state without evidence of disease at least 12 months after completing adjuvant or neoadjuvant hormonal therapy, as defined by 1 of the following:

    * PSA < 0.1 ng/mL after prostatectomy plus hormonal therapy
    * PSA < 0.5 ng/mL and has not doubled above nadir after radiotherapy plus hormonal therapy
  * Therapy lasted no more than 24 months
* Prior palliative radiotherapy allowed for participants, if commenced within 30 days before starting androgen deprivation.
* Bicalutamide, nilutamide or flutamide are allowed as single-agent therapy ≤ 28 days before medical castration to prevent flare.

Exclusion Criteria:

* PSA met criteria for PSA progression
* History of malignancy in the past 5 years, with the exception of basal cell and squamous cell carcinoma of the skin.
* Had any of the following within 6 months before randomization: myocardial infarction, severe/unstable angina pectoris, congestive heart failure, hospitalization for any cardiac event, including conduction abnormalities
* Pathological finding consistent with small cell, or neuroendocrine carcinoma of the prostate
* Known brain/ leptomeningeal metastases
* An active viral hepatitis (defined as Hepatitis B surface antigen [HBsAg] reactive or detectable [qualitative] HBV DNA defined as HCV Ribonucleic Acid [RNA] [qualitative] is detected), known human immunodeficiency virus infection with detectable viral load, or chronic liver disease with a need of treatment
* Uncontrolled hypertension as indicated by a resting systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite medical management
* A gastrointestinal (GI) disorder or procedure which is expected to interfere significantly with absorption of study drug
* Any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the participant and/or his compliance with study procedures or may interfere with the participant's participation in the study or evaluation of the study results.
* Prior hormone therapy in the metastatic setting
* Prior chemotherapy in the adjuvant or neoadjuvant setting
* Concurrent use or previous exposure of 5-alpha reductase inhibitors (within 28 days before the start of darolutamide or 5 half-lives of the drug, whichever is longer)
* Any Prior treatment with second-generation androgen receptor (AR) inhibitors such as enzalutamide, apalutamide, darolutamide, or other investigational AR inhibitors, Cytochrome P17 enzyme inhibitor such as abiraterone acetate or other investigational CYP 17 as antineoplastic treatment for prostate cancer
* Previous (within 28 days before the start of darolutamide or 5 half-lives of the investigational treatment of the previous study, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s).
* Contraindication to both CT and MRI contrast agent
* Hypersensitivity to any of the study treatments, study treatment classes, or excipients in the formulation of the study treatments
* Inability to swallow oral medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 12 months after end of enrollment
  Time interval from enrollment to PSA progression, clinical progression or death, whichever occurs first. PSA progression is defined as when the PSA demonstrates an increase that is more than 50% of nadir, taking as reference the lowest recorded PSA level since starting androgen deprivation therapy (ADT). Clinical progression is defined as increasing symptomatic bone metastases, radiographic progression per Response Evaluation Criteria In Solid Tumors (RECIST) criteria (v. 1.1) for soft tissue metastases and PCWG3 criteria for bone metastases, or clinical deterioration due to cancer per investigator's opinion.

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 24 months after end of enrollment
  Time from the date of enrollment until death resulting from any cause or the date last known alive
Radiographic Progression-free survival (rPFS) | Approximately 24 months after end of enrollment
  Time from enrollment to investigator-assessed radiographic progression per Response Evaluation Criteria In Solid Tumors (RECIST) criteria (v. 1.1) for soft tissue metastases and PCWG3 criteria for bone metastases or death, whichever occurs first
Time to castration-resistant prostate cancer (CRPC) | Approximately 12 months after end of enrollment
  Time from enrollment until documented clinical or PSA progression with a testosterone level of less than 50 ng per deciliter or documented medical castration or surgical castration
Complete PSA response rate | At 6 months after first administration
  PSA level of less than 0.2 ng per milliliter on two consecutive measurements at least 4 weeks apart
Number of participants with adverse events | From the signing of the informed consent form (ICF) until 30 (+7) days after last administration, approximately 12 months
  Adverse Events will be assessed by National Cancer Institute-Common Terminology Criteria (NCI CTCAE) v. 5.0

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Urology Centers of Alabama, PC - Homewood, Homewood, Alabama
  - Arizona Urology Specialists - Tucson - W Orange Grove, Tucson, Arizona
  - Tower Urology, Los Angeles, California
  - UCI Health Center for Urological Care, Orange, California
  - UC San Diego Health - Moores Cancer Center, San Diego, California
  - Providence Saint John's Cancer Institute, Santa Monica, California
  - Brigham and Women's Hospital (BWH) - Surgery Urology, Atlanta, Georgia
  - Piedmont Cancer Institute - Atlanta, Atlanta, Georgia
  - Northwestern Medicine - Urology, Chicago, Illinois
  - Northwestern University's Feinberg School of Medicine, Chicago, Illinois
  - UM Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Lieutenant Colonel Charles S. Kettles VA Medical Center - Oncology, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute - Detroit Headquarters, Detroit, Michigan
  - Michigan Institute of Urology - Troy - Town Center Building, Troy, Michigan
  - AMR - Kansas City, Kansas City, Missouri
  - GU Research Network, LLC - Oncology radiology, Omaha, Nebraska
  - XCancer Omaha, Omaha, Nebraska
  - New Jersey Urology - Clifton, Clifton, New Jersey
  - New Jersey Urology - Voorhees, Voorhees Township, New Jersey
  - New Mexico Cancer Center - Albuquerque, Albuquerque, New Mexico
  - Mount Sinai Doctors - Faculty Practice, New York, New York
  - Mount Sinai Faculty Practice Associates, New York, New York
  - Associated Medical Professionals of NY Syracuse, Syracuse, New York
  - The Urology Group - Norwood Surgery Center, Cincinnati, Ohio
  - Columbus Prostate Cancer Center / Radiation Oncology Clinic, Gahanna, Ohio
  - MidLantic Urology - Bala Cynwyd, Bala-Cynwyd, Pennsylvania
  - Carolina Urological Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC - Nashville, Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - Inova Schar Cancer Institute (vendor), Fairfax, Virginia
  - Spokane Urology PS, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] McKay RR, Ross AE, Preston MA, Gregg JR, Salami SS, Littleton N, Constantinovici N, Srinivasan S, Verholen F, Shore ND. Darolutamide plus androgen-deprivation therapy: propensity score matching of ARASEC and historic clinical trial patients. Future Oncol. 2025 May;21(11):1365-1375. doi: 10.1080/14796694.2025.2482360. Epub 2025 Apr 1. PMID 40165634
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21516